CLINICAL TRIAL: NCT05680428
Title: Effectiveness of Early Feeding Versus Conventional Feeding After Stoma Reversal in Adult Surgical Surgical Practices
Brief Title: Early Feeding Versus Conventional Feeding
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: DHQ mardan (Other)
Collaborators: DHQ HOSPITAL MARDAN (Unknown)
Responsible Party: Principal Investigator, Sajid Ali,FCPS, consultant General Surgeon, DHQ mardan
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 278-41
Record Dates: First submitted 2022-12-26; First posted 2023-01-11 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: Ileostomy - Stoma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- early feeding group (Experimental): after stoma reversal in patients in this group oral feeding was started with in 12 hrs after surgery
  Interventions: Other: early feeding
- conventional feeding group (Active Comparator): after stoma reversal in patients in this group oral feeding was started 48hrs after surgery
  Interventions: Procedure: conventional feeding

INTERVENTIONS:
Other: early feeding — oral feeding within 12hours after stoma reversal
  Arms: early feeding group
Procedure: conventional feeding — oral feeding after 48hours of NBM after stoma reversal
  Arms: conventional feeding group

SUMMARY:
The goal of this clinical trial is to compare early feeding vs conventional feeding after stoma reversal. The main question it aims to answer are:

• whether it is beneficial to start oral feeding within 12hrs after stoma reversal

Participants will be randomly assigned two groups either early feeding or conventional group

ELIGIBILITY:
Inclusion Criteria:

* having ileostomy
* no peritonitis
* intestinal obstruction

Exclusion Criteria:

* uncontrolled diabetes
* uncontrolled hypertension
* sepsis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2020-01-10 (Actual); Primary Completion 2022-06-10 (Actual); Study Completion 2022-07-10 (Actual)

PRIMARY OUTCOMES:
To evaluate the outcome of early versus conventional oral feeding in stoma reversal in terms of postoperative ileus | 5days
  comparison of post-op anastomotic leakage hospital stay wound infection

CONTACTS AND LOCATIONS:
Overall Officials: sajid khan, fcps, Principal Investigator — DHQ mardan
Locations (1):
- DHQ, Mardan, Kpk, Pakistan

IPD SHARING:
Plan to Share IPD: No